CLINICAL TRIAL: NCT03441789
Title: Efficacy and Safety of Enstilar Foam in Combination With Apremilast (Otezla) in Patients With Moderate Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: L.H. Kircik, M.D. (Other)
Responsible Party: Sponsor-Investigator, L.H. Kircik, M.D., Medical Director, Derm Research, PLLC
Organization: Derm Research, PLLC (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENS-1701
Record Dates: First submitted 2018-02-01; First posted 2018-02-22 (Actual); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — betamethasone dipropionate, calcipotriol drug combination; apremilast

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Otezla plus Enstilar foam (Experimental): Subjects randomized to this group will receive Otezla 30mg by mouth twice daily and Enstilar applied to affected areas once daily
  Interventions: Drug: Enstilar; Drug: Otezla
- Otezla plus vehicle foam (Placebo Comparator): Subjects in this group will take Otezla 30mg by mouth twice daily and vehicle foam applied to affected areas once daily
  Interventions: Drug: Vehicle; Drug: Otezla

INTERVENTIONS:
Drug: Enstilar — Enstilar foam applied to affected areas daily
  Other Names: calcipotriene and betamethasone dipropionate
  Arms: Otezla plus Enstilar foam
Drug: Vehicle — vehicle foam applied to affected areas once daily
  Arms: Otezla plus vehicle foam
Drug: Otezla — Otezla 30mg

SUMMARY:
This study seeks to show whether there is a benefit of prescribing Enstilar with Otezla in the treatment of patients with moderate plaque type psoriasis. Subjects will be randomized to study treatment at a 1:1 ratio of Otezla plus Enstilar foam versus Otezla plus vehicle foam.

DETAILED DESCRIPTION:
Approximately 50 subjects from 4 sites will be enrolled in this investigator-blind study. Subjects will be randomized 1:1 to Otezla plus Enstilar foam or Otezla plus vehicle foam and all adverse events and concomitant medications will be recorded.

Subjects will attend a screening visit/baseline visit and those with plaque-type psoriasis who have been started on commercial Otezla in the last 7 days will be randomized to study treatment as outlined above.

Enstilar or the vehicle will be initiated for the first 4 weeks and then Otezla will be continued as monotherapy for the next 8 weeks. Enstilar or the vehicle will be reinitiated for the last 4 weeks of the study. Total study period is 16 weeks and study visits will occur as follows: screening/baseline, week 1, 2, 3, 4, week 12, and week 16. Study assessments at each visit will be PASI, BSA, PGA, Itch VAS, DLQI, and standard medical assessments. There will be standard medication/treatment and washout periods.

ELIGIBILITY:
Inclusion Criteria:

I. Outpatient, male or female subjects of any race, 18 years of age or higher. Female subjects of childbearing potential must have a (-)UPT (urine pregnancy test) result at within 7 days of the first dose of study drug and practice a reliable method of contraception throughout the study;

A female is considered of childbearing potential unless she is:

- postmenopausal ≥ 5 years of age, without a uterus and/or both ovaries; or has been surgically sterile for ≥ 6 moths.

Reliable methods of contraception are:

- hormonal methods or IUD (intrauterine device) in use ≥ 90 days prior to study drug administration, barrier methods plus spermicide in use ≥ 14 days prior, or vasectomized partner.

[Exception: Female subjects of CBP (child bearing potential) who are not sexually active are not required to practice a reliable method of contraception and may be enrolled at the Investigator's discretion provided they are counseled to remain sexually inactive for the duration of the study and understand the risks involved in getting pregnant during the study.] ii. Subjects with moderate plaque type psoriasis who have been started on commercial Otezla within the last 10 days.

iii. Physician Global Assessment (PGA) score of 3. iv. Able to understand study requirements and sign Informed Consent/HIPAA forms.

Exclusion Criteria:

I. Female subjects who are pregnant, breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control, or male subjects planning a pregnancy with their spouse or partner while in the study.

ii. History of hypercalcemia or vitamin D toxicity or history of significant renal or hepatic disease iii. Patients with guttate, erythrodermic, or pustular psoriasis iv. Serious skin condition (other than psoriasis) or uncontrolled medical condition (in the opinion of the investigator).

v. Skin conditions (e.g.eczema) other than psoriasis that may interfere with evaluations of psoriasis.

vi. Known hypersensitivity to Enstilar Foam or any of its components. vii. Current drug or alcohol abuse (Investigator opinion). viii. Subject unable to commit to all the assessments required by the protocol. ix. Current enrollment in another clinical study and treatment with another experimental drug or approved therapy for experimental use within 30 days prior to the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Lawrence J. Green, MD LLC, Rockville, Maryland
  - Dermatology & Laser Center of Charleston, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant signed consent but failed screening
Period: Overall Study
Arm/Group | Otezla Plus Enstilar Foam | Otezla Plus Vehicle Foam
Started | 14 | 14
Completed | 13 | 10
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Otezla Plus Enstilar Foam: Subjects in the study will receive Otezla 30mg by mouth twice daily and Enstilar applied to affected areas once daily
  Enstilar: Enstilar foam applied to affected areas daily
  Otezla: Otezla 30mg
- Total: Total of all reporting groups
Arm/Group | Otezla Plus Enstilar Foam | Otezla Plus Vehicle Foam | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (17) | 52 (12) | 53 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With a Psoriasis Assessment and Severity Index (PASI) 75 at Week 16
Description: PASI combines the assessment of the severity of lesions and the area affected into a single score ranging from 0(no disease) to 72(maximal disease.) The body is divided into 4 sections: head (10% of total body surface area,) arms (20%,) trunk(30%,) and legs (40%.) Each of these is scored by itself and the 4 scores then combined to obtain thePASI. For each body area, the percent of skin area involved is estimated and graded based on this value (0=0% of area involved, 1=<10%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89%, 6=90-100%.) Within each area, the severity of disease is based on 3 clinical signs: erythema or redness, induration or thickness, and desquamation or scaliness. Each is graded on a scale from 0(none) to 4(maximum.) The sum of all 3 parameters is calculated for each body section, multiplied by the area score for that section and then multiplied by the weight of that section (.1for head, .2 arms, .3 trunk and .4 legs)
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Otezla Plus Enstilar Foam | Otezla Plus Vehicle Foam
Number analyzed (Participants) | 14 | 14
Participants | 7 | 2

2. Secondary Outcome: Percent of Subjects With PASI 75 at Week 4 and Week 12
Description: Psoriasis Area & Severity Index (PASI) is a tool used to measure the severity of psoriasis. It combines the assessment of the severity of lesions and the area affected into a single score ranging from 0(no disease) to 72(maximal disease.)
Time Frame: 4 weeks, 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Otezla Plus Enstilar Foam | Otezla Plus Vehicle Foam
Number analyzed (Participants) | 14 | 14
Participants
  week 4 | 7 | 1
  week 12 | 4 | 2

3. Secondary Outcome: Percent of Subjects With PASI 90 and 100 at Week 16
Description: as for outcome 2
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Otezla Plus Enstilar Foam | Otezla Plus Vehicle Foam
Number analyzed (Participants) | 14 | 14
Participants
  PASI 90 | 4 | 2
  PASI 100 | 1 | 0

4. Secondary Outcome: Per Cent of Patients With at Least 1-grade Improvement in Physicians Global Assessment (PGA) at Week 4 and Week 12 and Week 16
Description: The Investigator will rate the severity of of disease based on the assessment of 3 clinical signs (erythema, induration, desquamation) wherein 0=no signs of psoriasis, 1=almost clear, 2=mild, 3=moderate, 4=severe
Time Frame: 4 weeks, 12 weeks, 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Otezla Plus Enstilar Foam | Otezla Plus Vehicle Foam
Number analyzed (Participants) | 14 | 14
Participants
  week 4: clear | 1 | 0
  week 4: almost clear | 5 | 1
  week 4: mild | 7 | 4
  week 4: moderate | 1 | 9
  week 4: severe | 0 | 0
  week 12: clear | 1 | 0
  week 12: almost clear | 1 | 3
  week 12: mild | 5 | 4
  week 12: moderate | 6 | 7
  week 12: severe | 1 | 0
  week 16: clear | 1 | 1
  week 16: almost clear | 8 | 1
  week 16: mild | 4 | 3
  week 16: moderate | 0 | 9
  week 16: severe | 1 | 0

5. Secondary Outcome: Global Improvement in Itch Visual Analogue Scale (VAS) at Week 4,12 and 16
Description: The Itch VAS (Visual Analog Scale) is completed by subjects wherein they are asked to rate the severity of their itching over the last 48 hours on a scale from 0 (no itching) to 10 (unbearable itching); low scores indicate a better outcome.
Time Frame: 4 weeks, 12 weeks, 16 weeks
Measure: Mean (Standard Deviation); unit: scale unit
Arm/Group | Otezla Plus Enstilar Foam | Otezla Plus Vehicle Foam
Number analyzed (Participants) | 14 | 14
scale unit
  week 4 | 2 (2) | 5 (3)
  week 12 | 4 (3) | 4 (3)
  week 16 | 3 (3) | 4 (3)

6. Secondary Outcome: Global Percent Improvement in Dermatologic Quality of Life Index (DLQI) at Week 4, 12, and 16
Description: The DLQI is a 10-question tool completed by subjects to ascertain the severity of disease based on the extent to which disease interferes with daily life. Each question is scored according to the response wherein Very Much =3, A lot=2, A little=1 and Not at all=0. The sum of all responses is then recorded on a scale from 0 to 30, lower scores indicating better quality of life.
Time Frame: 4 weeks, 12, weeks, 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Otezla Plus Enstilar Foam | Otezla Plus Vehicle Foam
Number analyzed (Participants) | 14 | 14
score on a scale
  week 4 | 2 (2) | 5 (4)
  week 12 | 5 (5) | 5 (4)
  week 16 | 3 (4) | 6 (6)

ADVERSE EVENTS:
Time Frame: screening to week 16
Arm/Group | Otezla Plus Enstilar Foam | Otezla Plus Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/14 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Otezla Plus Enstilar Foam (N=14) | Otezla Plus Vehicle Foam (N=14)
sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
shortness of air (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Otezla Plus Enstilar Foam (N=14) | Otezla Plus Vehicle Foam (N=14)
increased joint pain generalized (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — right upper arm
overactive bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
dyspnea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
fall at home (General disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 0 (0) | 1 (1)
compressed lumbar disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
right flank pain (General disorders) | 1 (1) | 0 (0)
nausea (General disorders) | 1 (1) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
right ankle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
right lower jaw pain (General disorders) | 0 (0) | 1 (1)
root canal (Surgical and medical procedures) | 0 (0) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
frequent muscle fasciculation right lower eyelid (General disorders) | 0 (0) | 1 (1)
sensation of fullness in neck (General disorders) | 0 (0) | 1 (1)
persistent lower extremity edema (Cardiac disorders) | 0 (0) | 1 (1)
abrasion right shin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
headache (General disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
generalized rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03441789/Prot_SAP_000.pdf